CLINICAL TRIAL: NCT02567617
Title: Polyphenol Supplementation Inhibits Physiological Increase of Prostaglandin E2 During Reproductive Period - A Randomized Clinical Trial
Brief Title: Polyphenols Supplementation on Prostaglandin E2 in Women - Randomized Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Ana Maria Arregui Zilio, nutricionista, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4547/12; U1111-1173-3333 (Other: UTN)
Record Dates: First submitted 2015-09-30; First posted 2015-10-05 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Inflammatory Disorder of the Cardiovascular System
Keywords: Polyphenols, Prostaglandin E2, hormonal contraceptives
MeSH Terms: interventions — Polyphenols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Active Comparator): Group receiving capsules with polyphenols.
  Interventions: Dietary Supplement: Polyphenols
- Placebo controlled group (Placebo Comparator): Group receiving capsules with starch.
  Interventions: Dietary Supplement: Placebo controlled

INTERVENTIONS:
Dietary Supplement: Polyphenols — Capsules with five substances (polyphenols) at a concentration of 3000mg per day
  Arms: Intervention group
Dietary Supplement: Placebo controlled — Starch capsules
  Arms: Placebo controlled group

SUMMARY:
The aim of this study was to evaluate the effect of polyphenol supplementation on plasma levels of prostaglandin E2 in women during the reproductive period.

DETAILED DESCRIPTION:
The effect of anti-inflammatory substances on the constriction of the fetal ductus arteriosus is well documented, but the anti-inflammatory property of polyphenols and their effect on the metabolism of prostaglandins are not established. Evidence indicates that foods rich in polyphenols consumed from the third trimester of pregnancy may interfere with anatomical and functional activity of the fetal heart, presumably by the action similar to anti-inflammatory drugs nonsteroidal, causing inhibitory effect on prostaglandin synthesis. Objective: The objective of this study was to evaluate the effect of polyphenol supplementation on plasma levels of prostaglandin E2 in women of childbearing age use of hormonal contraceptives. As secondary endpoints were also evaluated other markers of inflammation and oxidative stress. The selected women were randomized to receive capsules polyphenol at a concentration of 3000 mg / day or placebo capsules to be consumed daily for fifteen days. Was applied dietary recall to assess intake of polyphenols, measured height and weight and carried blood samples for prostaglandin analysis E2 (PGE2), high sensitive C-reactive protein, and urine for analysis of total polyphenols and F2 isoprostane (8 iso-PGF2a). Statistical analysis: The results will be expressed through absolute and relative frequencies and mean ± standard deviation (SD) or median and interquartile range. For analysis, Pearson correlation is used. To compare the means will be used Student's t test. The level of significance is 5%. Considering a 90% power, with absolute error margin of 5% in the present study, 13 patients were needed in each group.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 25 to 35
* Use of hormonal contraceptives
* Agreed to participate and signed the Informed Consent

Exclusion Criteria:

* Pregnant women
* Use of anti-inflammatory drugs
* Using supplementation of omega 3
* BMI higher than 30 kg / m²
* Previous diagnosis of diabetes mellitus, hypertension, dyslipidemia, malignancy or infection

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Prostaglandin E2 | Baseline; 15 days
  markers analyzed in plasma

SECONDARY OUTCOMES:
F2 isoprostane | Baseline; 15 days
  marker analyzed i urine

OTHER OUTCOMES:
High sensitive C reactive protein | Baseline; 15 days
  markers analyzed in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Zielinsky, cardiologist, Study Director — Instituto de Cardiologia do Rio Grande do Sul

REFERENCES:
- [Background] Zielinsky P, Piccoli AL Jr, Manica JL, Nicoloso LH, Vian I, Bender L, Pizzato P, Pizzato M, Swarowsky F, Barbisan C, Mello A, Garcia SC. Reversal of fetal ductal constriction after maternal restriction of polyphenol-rich foods: an open clinical trial. J Perinatol. 2012 Aug;32(8):574-9. doi: 10.1038/jp.2011.153. Epub 2011 Nov 3. PMID 22052330